CLINICAL TRIAL: NCT00536549
Title: Effect of Real Time Continuous Glucose Monitoring System on the Management of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Responsible Party: Sei Hyun Baik, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Korean Health 21 R & D Project
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Type 2 Diabetes
Keywords: Glucose monitoring system; life style intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Guardina RT monitoring
  Interventions: Device: Guardian RT
- B (Active Comparator)
  Interventions: Behavioral: Education about the self monitoring blood glucose

INTERVENTIONS:
Device: Guardian RT
  Arms: A
Behavioral: Education about the self monitoring blood glucose
  Arms: B

SUMMARY:
The purpose of this study is to determine whether the Guardian Continuous Glucose Monitoring System in the home setting is more useful than frequent self blood glucose monitoring with a view to modifying patient's diet and exercise habits or improvement self disease control efforts and at last glycemic control in patients with type 2 diabetes

DETAILED DESCRIPTION:
In diabetes management, compliance, disease awareness and empowerment of the patient play an important role and the immediate feedback on the effects of diet and exercise that the self monitoring blood glucose (SMBG) may provide, could enhance patient empowerment. Increased use of SMBG has been shown to be associated with improved medication compliance and better metabolic control by several studies. However, because of many factors, including pain and inconvenience, many diabetic patients do not accept frequent fingersticks for self blood glucose monitoring (SBGM) levels. In addition, the SBGM result gives the data for only a few seconds, without any information on glucose trends.

So we need new glucose monitoring method that could reflect glucose trends and glycemic excursion continuously because glucose monitoring still remains the cornerstone of evaluating the efficacy of therapy and motivating self disease control in subjects with diabetes.

Few studies have examined the effects of real time continuous glucose monitoring system targeting type 2 diabetes. So our goal is to determine whether the Guardian Continuous Glucose Monitoring System in the home setting is more useful than frequent self blood glucose monitoring with a view to modifying patient's diet and exercise habits or improvement self disease control efforts and at last glycemic control in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Group 1: HbA1c < 8% with a stable insulin or oral hypoglycemic agents (OHA) regimen for the prior 2 months with no plans to switch modality of insulin or OHA administration during the next 3months.
* Group 2: HbA1c >= 8% and the fasting blood glucose must be < 130 at the same time with a stable insulin or oral hypoglycemic agents (OHA) regimen for the prior 2 months with no plans to switch modality of insulin or OHA administration during the next 3months

Exclusion Criteria:

* Use of corticosteroids or hormone therapy within the last 6 months
* Presence of another chronic illness

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
HbA1c, fasting blood glucose level, weight change, blood pressure in the morning, lipid profiles | basline, 12weeks later

SECONDARY OUTCOMES:
three day diary meals and seven day physical activity diary | basline, 12 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Sei H Baik, MD, Principal Investigator — Division of Endocrinology and Metabolism, Department of Internal Medicine,Korea University College of Medicine
Locations (1):
- Division of Endocrinology and Metabolism, Department of Internal Medicine,Korea University College of Medicine, Seoul, South Korea